CLINICAL TRIAL: NCT04623866
Title: A Single Center Randomized Controlled Clinical Study on the Treatment of Children With Purpura Nephritis With Huaiqihuang Granules
Brief Title: Study on the Treatment of Children With Purpura Nephritis With Huaiqihuang Granules
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, The Children's Hospital of Zhejiang University School of Medicine, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CXPJJH12000003-202017
Record Dates: First submitted 2020-10-25; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Henoch Schönlein Purpura Nephritis
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaiqihuang Group (Active Comparator): Huaiqihuang granules 60g/1.73m2 bid 24 weeks
  Interventions: Drug: Huaiqinhuang
- Valsartan group (Active Comparator): Valsartan granules 80mg/1.73m2 based qd 24 weeks
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: Huaiqinhuang — Huaiqihuang granules are composed of Huaier fungus, Fructus lycii and Huangjing. Studies have shown that huaiqihuang treatment can reduce cytokines in children with purpura nephritis interleukins IL - 4, IL - 10 and the tumor necrosis factor alpha (TNF alpha) expression level, prompt huaiqihuang granule treating children allergic purpura nephritis can significantly improve the clinical curative effect, improve the level of cytokines and the patient's immune function, and does not increase the incidence of adverse reactions.
  Other Names: Huaiqihuang granules
  Arms: Huaiqihuang Group
Drug: valsartan — Valsartan granules 80mg/1.73m2 based qd 24 weeks
  Other Names: Valsartan capsule
  Arms: Valsartan group

SUMMARY:
About 20% children with allergic purpura develop nephritis syndrome or nephrotic syndrome, 1% to 7% to kidney failure or end-stage renal disease. Children with serious damage to health, significantly reduced quality of life and caused heavy economic burden to the family . As the pathogenesis of HSPN is complex, it is difficult to formulate an exact individualized treatment plan.

DETAILED DESCRIPTION:
Children of Purpura nephritis with moderate protenuria(24 hours urinary protein quantitative 0.5 ~ 1.0 1.73 g/m2 and 24 hours urinary protein amount of not more than 1.0 g) in this study was choosed as participatant, plan randomly into the group of 10 cases, treated with huaiqihuang particles and valsartan for 24 weeks to analyze the curative effect and clinical value of single drug therapy for children with purpura nephritis in reducing proteinuria, protecting renal function and promoting rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. For children diagnosed with purpura nephritis, the diagnostic criteria for purpura nephritis shall refer to the 2016 edition of Evidence-based Guideline for diagnosis and Treatment of Purpura Nephritis published by the Nephrology Group of The Chinese Medical Association Pediatrics Branch, specifically as follows: Hematuria and/or proteinuria occur within 6 months of the course of allergic purpura. The diagnostic criteria for hematuria and proteinuria are as follows: A. Hematuria: gross hematuria or ≥3 RBC/high-power field (HP) under 3 times of microscope within 1 week. B. Proteinuria: if meeting any of the following conditions: 3 routine urine tests within 1 week qualitatively indicate positive urine protein; 24h quantitative urine protein >150 mg or urine protein/creatinine (mg/mg)>0.2; Urinary microalbumin was higher than normal for 3 times within 1 week. Very few children in the acute course of allergic purpura 6 months later, recurrent purpura, hematuria and/or proteinuria for the first time, should be sought for renal biopsy, such as IgA mesangial mesangial proliferative glomerulonephritis, can still be diagnosed as purpura nephritis.
2. 24-hour urinary protein quantification of 0.5 to 1.0g/1.73m2, and the total amount does not exceed 1.0g (to be quantified in non-infectious conditions);
3. Age: 6-14 years old;
4. Normal renal function: eGFR≥90ml/min/1.73m2;
5. Other manifestations of allergic purpura: skin purpura, abdominal pain, blood stool and joint swelling and pain have been relieved, and the use of hormone or immunosuppressive agents has been stopped for 2 weeks.

Exclusion Criteria:

1. Abnormal ophthalmic examination (fundus, visual field, photosensitivity);
2. Combined with gross hematuria;
3. Serious diseases of the heart, liver and other important organs, as well as diseases of the blood and endocrine system;
4. Patients who are known to be allergic to any component of Locust and wolfberry yellow or ACEI/ARB;
5. Patients who have participated in other clinical trials within three months before enrollment;
6. The investigator judged that the patient was not fit to participate in the study;(7) renal purpura nephritis wear results indicate Ⅲ magnitude or hints chronic purpura nephritis.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
change of urinary protein | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  24-hour urinary protein quantitative, urinary microprotein
Change in renal function of the patients | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  blood chemistry
change of lymphocyte subsets | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  including Th1 cells, Th2 cells, Th17 cells, cytokines (IL-16, IL-10, IL-17, etc.)
change of immunoglobulin + complement | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  immunoglobulin + complement
change of urine red blood cells | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  red blood cells routine urine

SECONDARY OUTCOMES:
Change of blood pressure | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  blood pressure
change of BMI(Body Mass Index) | before Clinical trials; 1 month, 2 months, 3 months, 6 months after randomization
  calculated by dividing weight in kilograms by height in meters squared( kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Mao Jianhua, Study Chair — Children's Hospital, Zhejiang University School of Medicine
Locations (2):
- China (2):
  - The Children Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
We could not share data without patients' agreement